CLINICAL TRIAL: NCT06915545
Title: Study on the Safety and Efficacy of the Aortic Arch Single Branch Covered Stent System for Aortic Dissection Involving the Aortic Arch
Brief Title: Study on the Aortic Arch Single Branch Stent Graft System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P158CT(CN)-01
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-03

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aortic Arch Single Branch Covered Stent System (Experimental): Aortic Arch Single Branch Covered Stent System for Aortic Dissection Involving the Aortic Arch
  Interventions: Device: Aortic Arch Single Branch Covered Stent System

INTERVENTIONS:
Device: Aortic Arch Single Branch Covered Stent System — to Evaluate the Safety and Efficacy of the Aortic Arch Single Branch Covered Stent System for Aortic Dissection Involving the Aortic Arch

SUMMARY:
The objective of the study is to evaluate the Safety and Efficacy of Aortic Arch Single Branch Covered Stent System for Aortic Dissection Involving the Aortic Arch

DETAILED DESCRIPTION:
The physician shall strictly follow the clinical study protocol and shall not deviate from or substantially change the protocol. However, in case of emergency such as immediate risk to the subjects, which needs tobe eliminated immediately, it may be reported in written form afterwards. During the course of the study,documents such as amendments to the clinical study protocol and informed consent, requests for deviation,and resumption of the suspended clinical study shall be subject to the written approval of the Ethics Committee

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years, gender unrestricted.
* Patients are diagnosed with Stanford Type B aortic dissection and need revascularization of the left subclavian artery.
* Anatomical criteria:

  * The diameter range of the proximal aortic landing zone is 20-42 mm.
  * The length of the proximal aortic landing zone (the distance from the posterior edge of the left common carotid artery orifice to the first intimal tear) is ≥15 mm.
  * The distance between the left common carotid artery and the left subclavian artery is ≥5 mm.
  * The length of the left subclavian artery landing zone is ≥25 mm, and the diameter range of the landing zone is 5-15 mm.
  * Suitable access to the femoral artery, iliac artery, and upper limb artery.
* Patients understand the purpose of the study, volunteer to participate, and are willing to complete follow - up visits as required by the protocol.

Exclusion Criteria:

* Previously undergone endovascular interventional treatment involving the aortic arch, or having a history of aortic surgical repair surgery, which affects the implantation and evaluation of the single branched covered stent system of the aortic arch.
* Patients with severe stenosis, calcification, or mural thrombus in the stent anchoring area pose challenges. Such conditions may easily prevent covered stents from adhering to the vessel wall or affect stent patency.
* Infectious aortic diseases, giant cell arteritis, Marfan syndrome (or other hereditary connective tissue diseases).
* Patients with systemic or local infections that may increase the risk of infection of the endovascular graft.
* Patients who have received abdominal aortic surgical or endovascular interventional surgery within the past 3 months.
* Patients who have had a stroke attack (excluding transient ischemic attack, TIA) or myocardial infarction within the past 3 months.
* Patients known to be allergic to contrast agents, stent materials, and delivery device materials (referring to nitinol, Dacron, PTFE, nylon polymer materials).
* Patients known to have contraindications to anticoagulant and antiplatelet drugs.
* Patients intolerant to general anesthesia.
* Patients with severe abnormalities in liver, kidney, and cardiac function before the operation [Subjects with a serum creatinine level exceeding 150 μmol/L; Subjects with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding 5 times the upper limit of the normal value; Subjects with serum total bilirubin (STB) exceeding 2 times the upper limit of the normal value; Subjects with a left ventricular ejection fraction lower than 50% as indicated by echocardiography.].
* Patients whose expected lifespan is shorter than 1 year.
* Female patients who are planning to conceive, are currently pregnant, or are breastfeeding.
* Patients whom, in the researcher's judgment, are not appropriate candidates for endovascular treatment.
* Patients who have been involved in other clinical studies and have not withdrawn from or exited the respective study groups within the three months preceding the screening period of this present study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate for freedom from major adverse events (MAE) within 30 days postoperatively | pre-discharge up to 14 days and 30 days post-surgery
  Major adverse events refer to the occurrences of all-cause death, myocardial infarction, renal failure, liver failure, respiratory failure, paraplegia, ischemic stroke, intestinal necrosis. Among them, renal failure means that it leads to persistent dialysis, kidney transplantation, or other fatal outcomes. Respiratory failure means that it leads to a significantly prolonged intubation time, tracheotomy, deterioration of lung function, or other fatal outcomes. Intestinal necrosis refers to intestinal ischemia that requires intestinal resection or leads to other fatal outcomes.
Procedural success rate of aortic dissection treatment 12 months postoperatively | intraoperative and 12 months postoperatively
  The composite endpoints include immediate technical success post-procedure and, at the 12-month CTA reexamination, the absence of displacement of the main aortic and branch stents, no type I or III endoleaks, patency of the branch stents, and no secondary surgical interventions during follow-up.

SECONDARY OUTCOMES:
All-cause mortality | Pre-discharge up to 14 days, 30 days post-surgery, 6 and 12 months and 2-5 years postoperatively
  All-cause mortality Refers to deaths from any cause that occur within the follow-up time points.
Mortality rate related to aortic dissection | Pre-discharge up to 14 days, 30 days post-surgery, 6 and 12 months and 2-5 years postoperatively
  Mortality rate related to aortic dissection refers to the death caused by the rupture of aortic dissection or the endovascular treatment of aortic dissection.
Incidence rate of severe adverse events | Pre-discharge up to 14 days, 30 days post-surgery, 6 and 12 months and 2-5 years postoperatively
  Serious adverse events refer to those occurring during the process of a clinical trial that lead to death or a serious deterioration of the health condition. This includes fatal diseases or injuries, permanent defects in body structures or body functions, the need for hospitalization or an extended hospital stay, and the requirement for medical or surgical interventions to prevent permanent defects in body structures or body functions.
Incidence rate of Device-related adverse events | Pre-discharge up to 14 days, 30 days post-surgery, 6 and 12 months and 2-5 years postoperatively
  Adverse events refer to adverse medical events that occur during the process of a clinical trial, regardless of whether they are related to the medical device used in the trial. However, normal postoperative stress responses should be distinguished, such as fever, discomfort in the chest and back, etc. If, upon the judgment of the researcher, it is determined to be a normal postoperative stress response, there is no need to record it as an adverse event of the medical device. Adverse events related to the medical device refer to situations that are determined by the researcher to be definitely related, possibly related, or undeterminable in relation to the medical device used in the trial.
The incidence rate of left upper limb ischemia | Pre-discharge up to 14 days, 30 days post-surgery, 6 and 12 months and 2-5 years postoperatively
  Left upper limb ischemia may present with weakness, coldness, pain, and numbness in the left upper limb. The ulnar artery, radial artery, and brachial artery may show weakened or absent pulsation.
Incidence rate of Type I/III endoleak | Intraoperative, pre-discharge（up to 14 days）, within 30 days and 6 and 12 months postoperatively
  A Type I endoleak occurs when there is a gap between the graft and the vessel wall at the "seal zones." This gap allows blood to flow alongside the graft into the aneurysm sac, creating pressure within the sac and increasing the risk of rupture. Type I endoleaks often occur when the aneurysm's anatomy is unsuitable for endovascular aneurysm repair (EVAR) or due to inappropriate device selection. However, vessel dilation over time can also cause this type of endoleak. Immediate attention is typically required because of the high risk of sac enlargement and rupture.
Incidence rate of stent graft migration | 6 and 12 months postoperatively
  Migration is defined as the single branched covered stent system of the aortic arch having a displacement of more than 10 mm compared with its position before discharge .
The patency rate of the branch vessel | Pre-discharge up to 14 days, 6 and 12 months postoperatively
  Branch vessel patency is defined as stenosis of ≤50%
The success rate of vascular remodeling for aortic dissection | within 30 days and 6 and 12 months postoperatively
  Evaluate the expansion of the true lumen and the thrombosis of the false lumen at the sites covered by the vascular stents for aortic dissection, so as to determine whether the vascular remodeling is successful.
The incidence rate of conversion to thoracotomy or secondary interventional surgery due to aortic dissection | Pre-discharge up to 14 days, 30 days post-surgery, 6 and 12 months and 2-5 years postoperatively
  Evaluate whether the subjects have been converted to thoracotomy or secondary interventional surgery due to aortic dissection.

CONTACTS AND LOCATIONS:
Overall Officials: chang shu, Professor, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Second Xiangya Hospital of Central South University, Changsha, China

IPD SHARING:
Plan to Share IPD: No